CLINICAL TRIAL: NCT00003178
Title: Idarubicin and Cladribine in Recurrent and Refractory Acute Myeloid Leukemia: A POG Phase II Study
Brief Title: Chemotherapy in Treating Children With Recurrent Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9720; COG-P9720 (Other: Children's Oncology Group); POG-9720 (Other: Pediatric Oncology Group); CDR0000065993 (Other: Clinical Trials.gov)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute promyelocytic leukemia (M3); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cladribine; 2'-chloro-2'-deoxyadenosine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1st Untreated Relapse for AML (Experimental): Patients receive idarubicin IV over 15 minutes on days 1-3, cladribine IV over 2 hours on days 1-5, and filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until blood counts have recovered for 2 days. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response after completion of course 1 may proceed to other chemotherapy or bone marrow transplantation at the discretion of the protocol investigator. Patients with extramedullary disease may receive intrathecal chemotherapy or radiotherapy to symptomatic sites.
  Interventions: Biological: filgrastim; Drug: cladribine; Drug: idarubicin
- Primary Refractory AML (Experimental): Patients receive idarubicin IV over 15 minutes on days 1-3, cladribine IV over 2 hours on days 1-5, and filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until blood counts have recovered for 2 days. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response after completion of course 1 may proceed to other chemotherapy or bone marrow transplantation at the discretion of the protocol investigator. Patients with extramedullary disease may receive intrathecal chemotherapy or radiotherapy to symptomatic sites.
  Interventions: Biological: filgrastim; Drug: cladribine; Drug: idarubicin
- MDS (Experimental): Patients receive idarubicin IV over 15 minutes on days 1-3, cladribine IV over 2 hours on days 1-5, and filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until blood counts have recovered for 2 days. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response after completion of course 1 may proceed to other chemotherapy or bone marrow transplantation at the discretion of the protocol investigator. Patients with extramedullary disease may receive intrathecal chemotherapy or radiotherapy to symptomatic sites.
  Interventions: Biological: filgrastim; Drug: cladribine; Drug: idarubicin

INTERVENTIONS:
Biological: filgrastim
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen®; NSC #614629
Drug: cladribine
  Other Names: 2-chlorodeoxyadenosine; CDA; Leustatin; NSC #105014)
Drug: idarubicin
  Other Names: 4-demethoxydaunorubicin; Idamycin; NSC#256439)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of idarubicin and cladribine in treating children who have recurrent acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete response rate in children with primary refractory or recurrent acute myeloid leukemia (AML) or secondary AML treated with idarubicin and cladribine. (Refractory AML stratum closed as of 4/3/01) (Secondary AML stratum closed as of 04/02/02)
* Compare the remission reinduction rates in children who relapse at 1 year or earlier vs more than 1 year from time of initial remission.
* Determine the toxic effects of this regimen in this patient population.

OUTLINE: Patients are stratified according to disease characteristics (primary or secondary acute myeloid leukemia (AML) with first untreated relapse vs primary refractory AML). (Refractory AML stratum closed as of 4/3/01) (Secondary AML stratum closed as of 04/02/02)

Patients receive idarubicin IV over 15 minutes on days 1-3, cladribine IV over 2 hours on days 1-5, and filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until blood counts have recovered for 2 days. Treatment repeats every 3 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response after completion of course 1 may proceed to other chemotherapy or bone marrow transplantation at the discretion of the protocol investigator. Patients with extramedullary disease may receive intrathecal chemotherapy or radiotherapy to symptomatic sites.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 51-102 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Acute myeloid leukemia (AML) (FAB M0-M7)
  * Secondary AML in first relapse (Secondary AML stratum closed as of 04/02/02)
  * AML in primary induction failure (Refractory AML stratum closed as of 04/03/01)
  * Myelodysplastic syndromes (MDS) (not related to Down syndrome) (MDS stratum closed as of 04/03/01)
* Extramedullary disease allowed
* Relapse more than 6 months after allogeneic or autologous bone marrow transplantation allowed

PATIENT CHARACTERISTICS:

Age:

* Under 21 at diagnosis

Performance status:

* Karnofsky 50-100% (over 10 years)
* Lansky 50-100% (10 years and under)

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 1.5 mg/dL
* ALT less than 3 times normal

Renal:

* Creatinine less than 2 times normal

Cardiovascular:

* Shortening fraction greater than 29%
* Ejection fraction greater than 55% with normal wall motion

Other:

* No uncontrolled infection
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* At least 12 weeks since prior idarubicin and recovered
* At least 2 weeks since other prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 1998-03; Primary Completion 2004-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival
  EFS will be estimated by Kaplan-Meier31 method. Prognostic factor analyses will be performed descriptively due to the limited sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Hurwitz, MD, Study Chair — Maine Children's Cancer Program at Barbara Bush Children's Hospital
Locations (235):
- United States (206):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Childhood Hematology/Oncology Associates, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami-Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Inc., Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Raymond Blank Memorial Hospital for Children, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's/Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - State University of New York Health Science Center at Brooklyn College of Medicine, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at JCMC, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Health Care System, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Charleston, Charleston, West Virginia
  - Cabell-Huntington Hospital, Inc, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Result] Chaleff S, Hurwitz CA, Chang M, Dahl G, Alonzo TA, Weinstein H. Phase II study of 2-chlorodeoxyadenosine plus idarubicin for children with acute myeloid leukaemia in first relapse: a paediatric oncology group study. Br J Haematol. 2012 Mar;156(5):649-55. doi: 10.1111/j.1365-2141.2011.08976.x. PMID 22512017